CLINICAL TRIAL: NCT02026128
Title: Objective Grading of Intraocular Inflammation in Uveitis Using Optical Coherence Tomography
Brief Title: Optical Coherence Tomography (OCT) in Uveitis
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, David Huang, MD, PhD, Professor of Ophthalmology & Director of Research, Casey Eye Institute OHSU, Oregon Health and Science University
Other Study IDs: OHSU IRB#00008052
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Uveitis
Keywords: Uveitis; Inflammation; OCT; Grading
MeSH Terms: conditions — Uveitis; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Active Uveitis: Physician-confirmed diagnosis of uveitis of any origin.

SUMMARY:
Optical Coherence Tomography (OCT) machines are non-contact instruments that can provide micrometer (one one-thousandths) scale imaging of biological tissue. This allows excellent assessment of the white blood and inflammatory cells seen in uveitis, an inflammation of any or all parts of the uvea (iris, ciliary body, choroid).

DETAILED DESCRIPTION:
In uveitis, white blood and inflammatory cells can enter the anterior chamber of the eye and adhere to the back surface of the cornea or enter the space between the lens and the retina in various types of uveitis. Transparency of the clear fluid that fills the space between the cornea and the lens (or between the lens and the retina) can be reduced due to the inflammation reaction of the eye. The amounts of these cells and reduced transparency that are present indicate the level of severity of inflammation.

The primary goal of this study is to use OCT to standardize anterior chamber (AC) cell grading. Another goal is to discover whether the size of cells and particles in the AC measured by OCT differs between uveitis diagnostic categories. OCT will also be used to detect protein concentration increases within the clear fluid inside the eye and determine if the concentration increase correlates with findings from the usual slit lamp grading method.

Background data including age, sex, medical history, and eye history will be gathered prior to the study/OCT testing visit. Other standard-of-care testing, like visual acuity and slit lamp (biomicroscope) exam will be performed to see if there is evidence of uveitis that meets the inclusion criteria for this study. If so, grading of the eye inflammation will be performed as defined by the Standardization of Uveitis Nomenclature (SUN). Once enrolled in the study, subjects will then undergo OCT testing with the study device to assess AC cells, AC flare (increased protein), keratic precipitates (cells adhered to back surface of cornea), and vitreous cells & haze (increased opacities in vitreous gel).

OCT Procedure: The subject will be seated and have their head positioned on a chin rest. They will be asked to look at a target (a lighted spot) while a beam of light scans the front part of the eye. The light is infrared and will not be visible or cause any sensation. A cotton tip swab may be used to help hold the eyelid open temporarily if necessary.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* With one or more of the following clinical features:

  1. >1+ AC cells;
  2. >1+ vitreous haze;
  3. presence of vitreous cells;
  4. presence of blood in anterior chamber;
  5. presence of blood in vitreous;
  6. presence of aqueous or vitreous pigment.
* In one of the following diagnostic categories as determined by a uveitis specialists:

  1. uveitis due to ankylosing spondylitis (positive HLA B27 genotype);
  2. uveitis due to sarcoidosis;
  3. uveitis of any additional type;
  4. uveitis masquerade such as pigment dispersion syndrome or Schaffer's sign;
  5. hyphema due to trauma or other causes;
  6. vitreous hemorrhage;
  7. retinal tear.

Exclusion Criteria:

* Inability to give informed consent;
* Inability to maintain stable fixation for OCT imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll both males and females and include all ethnic and racial groups through clinical practices. The study will enroll subjects 18 years of age or older with physician-confirmed, active uveitis. A total of thirty subjects will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2012-03; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of anterior chamber cells | 1 month
  Anterior chamber cells will be identified from OCT images by computer algorithms. Anterior chamber cells will be measured in particles.
Number of keratic precipitates (KP) | 1 month
  KPs will be identified from OCT images by computer algorithms. KPs will be measured in particles.
Number of vitreous cells | 1 month
  Vitreous cells will be identified from OCT images by computer algorithms. Vitreous cells will be measured in particles.
Degree of anterior chamber flare | 1 month
  OCT signal of the aqueous humor will be analyzed and correlated with slit lamp grades on AC flare. AC flare will be measured in a.u.

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States